CLINICAL TRIAL: NCT03930485
Title: Risk Factors for Persistent Postural-Perceptual Dizziness Development
Acronym: RIPPPDD
Status: Completed | Type: Observational
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 09042019
Record Dates: First submitted 2019-04-09; First posted 2019-04-29 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Dizziness
MeSH Terms: conditions — Dizziness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of this study is to determine whether the prevalence of neuroticism, anxiety and body vigilance is higher in patients diagnosed with PPPD compared to those who suffered a vestibular insult but did not develop PPPD and healthy controls. An increased prevalence of one or more of these factors may identify them as risk factors in the development of PPPD. The secondary aim is to understand how PPPD affects quality of life.

DETAILED DESCRIPTION:
The diagnosis persistent postural-perceptual dizziness (PPPD) entered the 11th edition of the World Health Organization's International Classification of Diseases (ICD-11 beta draft) in 2015 following a consensus document on its diagnostic criteria created by the Behavioral Subcommittee of the Committee for the Classification of Vestibular Disorders of the Bárány Society (CCBS) between 2010 and 2014. The ICD-11 describes it as follows: "Persistent non-vertiginous dizziness, unsteadiness, or both lasting three months or more. Symptoms are present most days, often increasing throughout the day, but may wax and wane. Momentary flares may occur spontaneously or with sudden movement. Affected individuals feel worst when upright, exposed to moving or complex visual stimuli, and during active or passive head motion. These situations may not be equally provocative. Typically, the disorder follows occurrences of acute or episodic vestibular or balance-related problems, but may follow non-vestibular insults as well. Symptoms may begin intermittently, and then consolidate. Gradual onset is uncommon." In a previous systematic review of the literature, the authors discuss the pathophysiology and management of PPPD, including certain psychological risk factors. Anxiety has been suggested to play a pivotal role in the maladaptation cycle of PPPD in part by increasing body vigilance and both neuroticism and a pre-existing anxiety disorder have been suggested as predisposing factors for the onset of this maladaptation cycle. Such risk factors may allow the prediction of who might be at risk of developing PPPD after an acute vestibular injury and thus benefit from early treatment.

As PPPD is a relatively new diagnosis, to date there is no study that comprehensively confirms the prevalence of anxiety, neuroticism and/or increased body vigilance in sufferers specifically. It is important to determine this in order to guide further research into treating and potentially preventing its onset.

ELIGIBILITY:
Inclusion Criteria

* Must have diagnosis of PPPD based on the CCBS criteria
* Aged under 18 years old
* Able to provide informed consent Exclusion Criteria
* No confirmed/firm diagnosis of PPPD
* Aged <18 years old
* Unable to provide informed consent
* Current clinically significant illness that could confound the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have been given a previous diagnosis of PPPD will be considered as potential cases and screened for inclusion/exclusion criteria. PPPD diagnosis must be based on the CCBS criteria (Table 1). Participants will be identified by a member of the current clinical care team either through clinic notes or in the outpatient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Scores of the Generalised Anxiety & Depression - 7 (GAD-7) questionnaire | 1 year
  Average total scores of the GAD-7 will be compared across each study group. Higher scores indicate higher feelings of anxiety and/or depression in that study group. The minimum score is 0 and the maximum is 21.
Scores of the Big Five Inventory (BFI) questionnaire | 1 year
  Average total scores for each category of the BFI will be compared across each study group. The BFI measures five personality areas: Extraversion, Aggreableness, Conscientiousness, Neuroticism, and Openess. Minimum scores for each subcategory is 1 and the maximum is 5. Higher scores indicate a higher propensity for that personality trait.
Scores from the Body Vigilance Scale (BVS) questionnaire | 1 year
  Average scores for each question of the BVS will be compared across each study group. Minimum score is 0, maximum score is 10. Higher scores indicate higher body vigilance towards bodily sensations.

SECONDARY OUTCOMES:
Scores from the Dizziness Handicap Inventory (DHI) questionnaire | 1 year
  Average total scores for the DHI will be compared across each study group. Minimum score is 0, maximum is 50, higher scores indicate more symptoms of dizziness in day to day life.
Scores from the Vertigo Symptom Scale (VSS) questionnaire | 1 year
  Average total scores for the VSS will be compared across each study group. Minimum score is 0, maximum is 60. Higher scores indicate a higher severity of symptoms caused by vertigo.
Scores from the Brief Dizziness Perception Questionnaire (DPQ) | 1 year
  Average scores from each question of the DPQ will be measure across each study group. Minimum score is 0, maximum is 10. Higher scores indicate an individual is more affected/more concerned etc regarding their dizziness.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Trinidade, MBBS, Principal Investigator — CI; Bhaskar Dasgupta, MD, Study Director — R&D Director
Locations (1):
- Southend Hospital, Westcliff-on-Sea, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No